CLINICAL TRIAL: NCT01946074
Title: A Multicenter, Phase 1/1b, Open-Label, Dose-Escalation Study of ABT-165, a Dual Variable Domain Immunoglobulin in Subjects With Advanced Solid Tumors
Brief Title: A Study of ABT-165 in Subjects With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M14-006
Record Dates: First submitted 2013-09-17; First posted 2013-09-19 (Estimated); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Advanced Solid Tumors
Keywords: ABBV-181; ABT-165; cancer; neoplasm; advanced solid tumor; colorectal cancer
MeSH Terms: conditions — Neoplasms; Colorectal Neoplasms | interventions — Paclitaxel; IFL protocol; ABT-165; budigalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Monotherapy (Experimental): ABT-165 will be administered at escalating dose levels in 28-day dosing cycles (2 doses per cycle). Additional subjects will be enrolled in an expansion cohort that will further evaluate ABT-165
  Interventions: Drug: ABT-165
- Cohort A (Experimental): ABT-165 plus paclitaxel
  Interventions: Drug: paclitaxel; Drug: ABT-165
- Cohort B (Experimental): ABT-165 plus FOLFIRI
  Interventions: Drug: FOLFIRI; Drug: ABT-165
- Cohort C (Experimental): ABT-165 plus ABBV-181
  Interventions: Drug: ABT-165; Drug: ABBV-181
- Cohort D (Experimental): ABT-165 plus ABBV-181 plus paclitaxel
  Interventions: Drug: paclitaxel; Drug: ABT-165; Drug: ABBV-181

INTERVENTIONS:
Drug: paclitaxel — Paclitaxel will be administered by intravenous infusion.
  Arms: Cohort A; Cohort D
Drug: FOLFIRI — 5-fluorouracil, Folinic acid and Irinotecan will be administered by intravenous infusion.
  Arms: Cohort B
Drug: ABT-165 — ABT-165 will be administered by intravenous infusion at escalating dose levels.
Drug: ABBV-181 — ABBV-181 will be administered by intravenous infusion.
  Arms: Cohort C; Cohort D

SUMMARY:
This is a Phase 1/1b open-label study evaluating the safety, pharmacokinetics (PK), and preliminary efficacy of ABT-165 when administered as monotherapy and in combination with paclitaxel or 5-fluoruracil, folinic acid and irinotecan (FOLFIRI) or ABBV-181 with/without paclitaxel in subjects with advanced solid tumors. Enrollment to Cohorts A, B were completed and for Cohorts C and D are recruiting.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have advanced solid tumor that is not amenable to surgical resection or other approved therapeutic options that have demonstrated clinical benefit.
* Subject has adequate bone marrow, renal, hepatic and coagulation function.
* Subject must have measurable disease per Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1 or disease evaluable by assessment of tumor antigens including but not limited to cancer antigen (CA-125) and prostate-specific antigen (PSA).
* Women of childbearing potential must have a negative serum pregnancy test at the screening visit and a negative urine pregnancy test at baseline prior to the first dose of study drug. Female subject considered not of childbearing potential must be documented as being surgically sterile or post-menopausal for at least 1 year. Women of childbearing potential and men must agree to use adequate contraception.
* Subjects in the combination therapy cohorts must meet the above inclusion criteria and be eligible to receive paclitaxel or FOLFIRI per most current prescribing information, or at the discretion of the Investigator. Subjects in the combination therapy cohorts who are to receive ABBV-181, an anti-PD1 antibody, must also meet other criteria described in the Protocol.

Exclusion Criteria:

* Subject has received anticancer therapy including chemotherapy, radiation therapy, immunotherapy, biologic, or any investigational therapy within a period of 21 days or anti-cancer herbal therapy within 7 days prior to Cycle 1 Day 1 of ABT-165.
* Subject has uncontrolled metastases to the central nervous system (CNS).
* Subject has unresolved clinically significant toxicities from prior anticancer therapy, defined as any Common Terminology Criteria for Adverse Events (CTCAE) Grade 2 or higher.
* Subject has history (within previous 5 years) of clinically significant pulmonary hypertension, uncontrolled systemic hypertension or hypertensive crisis, symptomatic heart failure, cardiomyopathy, myocardial infarction, unstable/severe angina pectoris, cardiac arrhythmia requiring medication, coronary/peripheral artery bypass graft, aneurysm or aneurysm repair, angioplasty, cerebrovascular accident, transient ischemic attack or the left ventricular ejection fraction (LVEF) less than 50%.
* Subjects enrolled on the combination therapy phase must not meet the above exclusion criteria and must be eligible to receive paclitaxel or FOLFIRI per most current prescribing information, or at the discretion of the Investigator. Subjects receiving ABBV-181 must not meet other exclusion criteria described in the Protocol.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2013-08-08 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2022-09-28 (Actual)

PRIMARY OUTCOMES:
Clinical lab testing | Up to 30 days after a 24-month treatment period
  Hematology, Chemistry, and Urinalysis
Maximum observed serum concentration (Cmax) of ABT-165 | Up to 90 days after a 24-month of treatment period
The terminal elimination half life of ABT-165 | Up to 90 days after a 24-month treatment period
Cardiac assessment | Up to 30 days after a 24-month treatment period
  Electrocardiogram (ECG), echocardiogram (ECHO), basic natriuretic peptide (BNP) and troponin I
Area under the curve (AUC) form time zero to the last measurable concentration AUC (0-t) | Up to 90 days after a 24-month treatment period
  AUC (0-t) = Area under the serum concentration versus time curve form time zero (pre-dose) to the time of the last measurable concentration
Physical exam | Up to 30 days after a 24-month treatment period
  Assessment of normal/abnormal physical findings
Number of participants with Adverse Events | Up to 90 days after a 24-month treatment period
  Collect all adverse events at each visit
Vital signs | Up to 30 days after a 24-month treatment period
  Blood pressure, heart rate, respiratory rate and body temperature

SECONDARY OUTCOMES:
Duration of overall response (DOR) | Up to 30 days after a 24-month treatment period
  DOR is defined as the time from the subject's initial CR or PR to the time of disease progression
Objective response rate (ORR) | Up to 30 days after a 24-month treatment period
  ORR is defined as the proportion of the subjects who have a complete response (CR) or partial response (PR)
Progression free survival (PFS) | Up to 30 days after a 24-month treatment period
  PFS is defined as the time from the first dose date of ABT-165 to either disease progression or death, whichever occurs first

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (10):
- United States (10):
  - HonorHealth Research Institute - Pima /ID# 105677, Scottsdale, Arizona
  - Scottsdale Healthcare /ID# 105678, Scottsdale, Arizona
  - University of California, Los Angeles /ID# 141389, Los Angeles, California
  - University of California, Davis Comprehensive Cancer Center /ID# 141164, Sacramento, California
  - Stanford University School of Med /ID# 123758, Stanford, California
  - Illinois Cancer Care, PC /ID# 151970, Peoria, Illinois
  - Horizon Oncology Research Center /ID# 138022, Lafayette, Indiana
  - Duke Cancer Center /ID# 105679, Durham, North Carolina
  - Tennessee Oncology-Nashville Centennial /ID# 143280, Nashville, Tennessee
  - Mary Crowley Cancer Research /ID# 123757, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gordon MS, Nemunaitis J, Barve M, Wainberg ZA, Hamilton EP, Ramanathan RK, Sledge GW Jr, Yue H, Morgan-Lappe SE, Blaney M, Kasichayanula S, Motwani M, Wang L, Naumovski L, Strickler JH. Phase I Open-Label Study Evaluating the Safety, Pharmacokinetics, and Preliminary Efficacy of Dilpacimab in Patients with Advanced Solid Tumors. Mol Cancer Ther. 2021 Oct;20(10):1988-1995. doi: 10.1158/1535-7163.MCT-20-0985. Epub 2021 Jul 26. PMID 34315767